CLINICAL TRIAL: NCT02570321
Title: Cross-linking for Corneal Ulcers Treatment Trial
Acronym: CLAIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Aravind Eye Hospitals, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-14918
Record Dates: First submitted 2015-09-15; First posted 2015-10-07 (Estimated); Results first posted 2024-08-27 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Corneal Ulcer; Infectious Keratitis; Bacterial Ulcer; Fungal Ulcer
Keywords: Cornea; Ulcer; Infectious keratitis; Bacterial; Fungal
MeSH Terms: conditions — Corneal Ulcer; Corneal Diseases; Ulcer | interventions — Corneal Cross-Linking

STUDY DESIGN:
Intervention Model Description: Patients with corneal ulcers are randomized to topical antimicrobial plus corneal crosslinking versus topical antimicrobial alone
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Bacterial ulcer cross-linking (Experimental): Standard of care topical treatment for bacterial ulcer plus cross-linking
  Interventions: Procedure: Corneal Cross-linking
- Bacterial ulcer control (Active Comparator): Standard of care topical treatment for bacterial ulcer
  Interventions: Procedure: Corneal Cross-linking
- Fungal ulcer cross-linking plus natamycin (Experimental): Standard of care topical treatment for fungal ulcer with natamycin plus cross-linking
  Interventions: Procedure: Corneal Cross-linking; Drug: Anti Fungal Drug
- Fungal ulcer control with natamycin (Active Comparator): Standard of care topical treatment for fungal ulcer with natamycin
  Interventions: Procedure: Corneal Cross-linking; Drug: Anti Fungal Drug
- Fungal ulcer cross-linking plus amphotericin (Experimental): Standard of care topical treatment for fungal ulcer with amphotericin plus cross-linking
  Interventions: Procedure: Corneal Cross-linking; Drug: Anti Fungal Drug
- Fungal ulcer control with amphotericin (Active Comparator): Standard of care topical treatment for fungal ulcer with amphotericin
  Interventions: Procedure: Corneal Cross-linking; Drug: Anti Fungal Drug

INTERVENTIONS:
Procedure: Corneal Cross-linking — For those subjects randomized to receive collagen cross-linking, the procedure will be performed as per the routine at the hospital (UV-X machine; strict aseptic precautions; corneal epithelium debrided and 0.1% riboflavin applied for 30 minutes, then UV-A radiation applied for 30 minutes at 370nm with 3mW/cm2). Corneal cross-linking is a routine procedure performed by Aravind Eye Hospital for infectious keratitis.
Drug: Anti Fungal Drug — Topical Amphotericin B vs Topical Natamycin
  Arms: Fungal ulcer control with amphotericin; Fungal ulcer control with natamycin; Fungal ulcer cross-linking plus amphotericin; Fungal ulcer cross-linking plus natamycin

SUMMARY:
The primary purpose of this study is to determine if patients randomized to corneal collagen cross-linking plus medical therapy will have a lower prevalence of positive bacterial or fungal cultures immediately after the procedure than patients who received medical therapy alone.

The secondary purpose of this study is to determine if patients randomized to corneal collagen cross-linking will have a better visual acuity at 3 and 12 months than patients who receive medical therapy alone.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial to determine whether collagen cross-linking improves outcomes in microbial keratitis. Patients presenting to the Aravind Eye Hospitals in Madurai, India for treatment of microbial keratitis will be recruited for the proposed study. Approximately 266 patients will be enrolled in the study. Subjects presenting with bacterial keratitis will be randomized to receive medical therapy plus corneal collagen cross-linking at presentation or to receive medical therapy alone. All subjects with bacterial ulcers will receive standard topical antibiotic medications as required after the procedure.

Subjects with fungal keratitis will be randomized into one of four groups:

1. collagen cross-linking + amphotericin;
2. collagen cross-linking + natamycin;
3. amphotericin alone;
4. natamycin alone.

All study subjects will be followed for 12 months to evaluate response to treatment.

Investigators from the University of California, San Francisco (UCSF) will assist Aravind Eye Hospital with the study design, implementation, and analysis of the research, and will help fund the study. The investigators plan to visit Aravind to help with the study implementation. UCSF will play an important role in this study by assisting with the study design, implementation, analysis, and funding.

ELIGIBILITY:
Inclusion criteria:

* Corneal ulcer that is smear positive for either bacteria or filamentous fungus
* Pinhole visual acuity worse than 20/70 in the affected eye
* Not treated already with antimicrobial medications at presentation
* Age over 18 years
* Basic understanding of the study as determined by the physician
* Commitment to return for follow up visits

Exclusion criteria:

* Evidence of concomitant infection on exam or gram stain (i.e. herpes, both bacteria and acanthamoeba on gram stain)
* Impending or frank perforation at recruitment
* Involvement of sclera at presentation
* Non-infectious or autoimmune keratitis
* History of corneal transplantation or recent intraocular surgery
* No light perception in the affected eye
* Pinhole visual acuity worse than 20/200 in the unaffected eye
* Participants who are decisionally and/or cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Rose-Nussbaumer, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- Proctor Foundation, UCSF, San Francisco, California, United States
- Aravind Eye Hospitals, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prajna NV, Radhakrishnan N, Lalitha P, Liu Z, Keenan JD, Arnold BF, Rose-Nussbaumer J. Mediators of the Effect of Corneal Cross-Linking on Visual Acuity for Fungal Ulcers: A Prespecified Secondary Analysis From the Cross-Linking-Assisted Infection Reduction Trial. Cornea. 2022 Oct 1;41(10):1217-1221. doi: 10.1097/ICO.0000000000002965. Epub 2022 Jan 17. PMID 35044972
- [Derived] Prajna NV, Lalitha P, Krishnan T, Rajaraman R, Radnakrishnan N, Srinivasan M, Devi L, Das M, Liu Z, Zegans ME, Acharya NR, Porco TC, Lietman TM, Rose-Nussbaumer J. Patterns of Antifungal Resistance in Adult Patients With Fungal Keratitis in South India: A Post Hoc Analysis of 3 Randomized Clinical Trials. JAMA Ophthalmol. 2022 Feb 1;140(2):179-184. doi: 10.1001/jamaophthalmol.2021.5765. PMID 35024776
- [Derived] Prajna NV, Radhakrishnan N, Lalitha P, Rajaraman R, Narayana S, Austin AF, Liu Z, Keenan JD, Porco TC, Lietman TM, Rose-Nussbaumer J. Cross-Linking Assisted Infection Reduction (CLAIR): A Randomized Clinical Trial Evaluating the Effect of Adjuvant Cross-Linking on Bacterial Keratitis. Cornea. 2021 Jul 1;40(7):837-841. doi: 10.1097/ICO.0000000000002510. PMID 33079921
- [Derived] Prajna NV, Radhakrishnan N, Lalitha P, Austin A, Liu Z, Keenan JD, Porco TC, Lietman TM, Rose-Nussbaumer J. Cross-Linking Assisted Infection Reduction: One-year Follow-up of a Randomized Clinical Trial Evaluating Cross-Linking for Fungal Keratitis. Ophthalmology. 2021 Jun;128(6):950-952. doi: 10.1016/j.ophtha.2020.09.042. Epub 2020 Oct 5. No abstract available. PMID 33031809
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558
- [Derived] Prajna NV, Radhakrishnan N, Lalitha P, Austin A, Ray KJ, Keenan JD, Porco TC, Lietman TM, Rose-Nussbaumer J. Cross-Linking-Assisted Infection Reduction: A Randomized Clinical Trial Evaluating the Effect of Adjuvant Cross-Linking on Outcomes in Fungal Keratitis. Ophthalmology. 2020 Feb;127(2):159-166. doi: 10.1016/j.ophtha.2019.08.029. Epub 2019 Sep 4. PMID 31619359

RESULTS

PARTICIPANT FLOW:
Groups:
- Bacterial Ulcer Control: Standard of care topical treatment for bacterial ulcer
  Bacterial ulcer control: For those bacterial ulcer subjects randomized to the control group, they will receive the standard of care topical treatment for bacterial ulcers. This group will have their eyes irrigated with a balanced salt solution.
- Bacterial Ulcer Cross-linking: Standard of care topical treatment for bacterial ulcer plus cross-linking
  Bacterial ulcer cross-linking: For those subjects randomized to receive collagen cross-linking, the procedure will be performed as per the routine at the hospital (UV-X machine; strict aseptic precautions; corneal epithelium debrided and 0.1% riboflavin applied for 30 minutes, then UV-A radiation applied for 30 minutes at 370nm with 3mW/cm2). Corneal cross-linking is a routine procedure performed by Aravind Eye Hospital for infectious keratitis.
- Fungal Ulcer Control With Natamycin: Standard of care topical treatment for fungal ulcer with natamycin
  Fungal ulcer control: Prior to receiving sham cross-linking, topical amphotericin B or topical natamycin antifungal therapy will be started as per routine at the hospital; a loading dose of amphotericin B or natamycin every 5 minutes x 6 will be followed by dosing every 30 minutes. Amphotericin B and natamycin are routinely used therapies for fungal keratitis at Aravind Eye Hospital.
  For those fungal ulcer subjects randomized to the control group, they will receive the standard of care topical treatment for fungal ulcers. This group will have their eyes irrigated with a balanced salt solution.
- Fungal Ulcer Cross-linking Plus Natamycin: Standard of care topical treatment for fungal ulcer with natamycin plus cross-linking
  Fungal ulcer cross-linking: Prior to receiving cross-linking, topical amphotericin B or topical natamycin antifungal therapy will be started as per routine at the hospital; a loading dose of amphotericin B or natamycin every 5 minutes x 6 will be followed by dosing every 30 minutes. Amphotericin B and natamycin are routinely used therapies for fungal keratitis at Aravind Eye Hospital.
  For those subjects randomized to receive collagen cross-linking, the procedure will be performed as per the routine at the hospital (UV-X machine; strict aseptic precautions; corneal epithelium debrided and 0.1% riboflavin applied for 30 minutes, then UV-A radiation applied for 30 minutes at 370nm with 3mW/cm2). Corneal cross-linking is a routine procedure performed by Aravind Eye Hospital for infectious keratitis.
- Fungal Ulcer Control With Amphotericin: Standard of care topical treatment for fungal ulcer with amphotericin
  Fungal ulcer control: Prior to receiving sham cross-linking, topical amphotericin B or topical natamycin antifungal therapy will be started as per routine at the hospital; a loading dose of amphotericin B or natamycin every 5 minutes x 6 will be followed by dosing every 30 minutes. Amphotericin B and natamycin are routinely used therapies for fungal keratitis at Aravind Eye Hospital.
  For those fungal ulcer subjects randomized to the control group, they will receive the standard of care topical treatment for fungal ulcers. This group will have their eyes irrigated with a balanced salt solution.
- Fungal Ulcer Cross-linking Plus Amphotericin: Standard of care topical treatment for fungal ulcer with amphotericin plus cross-linking
  Fungal ulcer cross-linking: Prior to receiving cross-linking, topical amphotericin B or topical natamycin antifungal therapy will be started as per routine at the hospital; a loading dose of amphotericin B or natamycin every 5 minutes x 6 will be followed by dosing every 30 minutes. Amphotericin B and natamycin are routinely used therapies for fungal keratitis at Aravind Eye Hospital.
  For those subjects randomized to receive collagen cross-linking, the procedure will be performed as per the routine at the hospital (UV-X machine; strict aseptic precautions; corneal epithelium debrided and 0.1% riboflavin applied for 30 minutes, then UV-A radiation applied for 30 minutes at 370nm with 3mW/cm2). Corneal cross-linking is a routine procedure performed by Aravind Eye Hospital for infectious keratitis.
Period: Overall Study
Arm/Group | Bacterial Ulcer Control | Bacterial Ulcer Cross-linking | Fungal Ulcer Control With Natamycin | Fungal Ulcer Cross-linking Plus Natamycin | Fungal Ulcer Control With Amphotericin | Fungal Ulcer Cross-linking Plus Amphotericin
Started | 19 | 17 | 26 | 27 | 30 | 28
Completed | 17 | 16 | 21 | 27 | 27 | 25
Not Completed | 2 | 1 | 5 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bacterial Ulcer Control | Bacterial Ulcer Cross-linking | Fungal Ulcer Control With Natamycin | Fungal Ulcer Cross-linking Plus Natamycin | Fungal Ulcer Control With Amphotericin | Fungal Ulcer Cross-linking Plus Amphotericin | Total
Number analyzed (Participants) | 19 | 17 | 26 | 27 | 30 | 28 | 147
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [54.5 to 65] | 59 [48 to 66] | 50 [36 to 55] | 55 [47 to 65] | 45 [40 to 58] | 56 [45 to 65] | 54.5 [45 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 9 | 12 | 16 | 11 | 63
  Male | 13 | 8 | 17 | 15 | 14 | 17 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 19 | 17 | 26 | 27 | 30 | 28 | 147
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  India | 19 | 17 | 26 | 27 | 30 | 28 | 147
Occupation [Count of Participants; unit: Participants]
  Agriculture | 12 | 8 | 16 | 13 | 18 | 13 | 80
  Nonagriculture | 6 | 9 | 10 | 14 | 12 | 15 | 66
  NA | 1 | 0 | 0 | 0 | 0 | 0 | 1
Medication use at enrollment [Count of Participants; unit: Participants] | 8 | 10 | 18 | 21 | 19 | 24 | 100
Affected Eye [Count of Participants; unit: Participants]
  Left | 8 | 8 | 11 | 12 | 18 | 13 | 70
  Right | 11 | 9 | 15 | 15 | 12 | 15 | 77
Visual acuity [Mean (Inter-Quartile Range); unit: LogMar] — Uncorrected and pinhole visual acuity will be measured at baseline for both eyes using the standard ETDRS chart light box at the 4- and 1-meter test distances. In the case that the patient reads less than 10 letters at 4 meters, move the patient or the chart to a distance of 1 meter from the patient.
  LogMar | 1.7 [0.7 to 1.7] | 1.7 [0.9 to 1.8] | 1.05 [0.62 to 1.12] | 1.1 [0.6 to 1.7] | 1.05 [0.62 to 1.7] | 1.22 [0.91 to 1.7] | 1.1 [0.63 to 1.7]
Ulcer location [Count of Participants; unit: Participants]
  Central | 14 | 13 | 21 | 23 | 26 | 22 | 119
  Peripheral | 4 | 4 | 5 | 4 | 4 | 6 | 27
  NA | 1 | 0 | 0 | 0 | 0 | 0 | 1
Infiltrate and/or scar [Mean (Inter-Quartile Range); unit: mm] | 3.5 [2.7 to 4] | 3 [2.24 to 4] | 3.0 [2.5 to 3.5] | 3.9 [2.6 to 4.5] | 3.5 [2.7 to 4.5] | 3.1 [2.8 to 5.0] | 3.3 [2.5 to 4.5]
Hypopyon [Count of Participants; unit: Participants]
  No | 6 | 6 | 19 | 16 | 15 | 14 | 76
  <0.5 mm | 2 | 1 | 1 | 5 | 5 | 1 | 15
  >=0.5 mm | 11 | 10 | 6 | 6 | 10 | 13 | 56
% Depth [Count of Participants; unit: Participants]
  >0-33% | 5 | 6 | 14 | 13 | 13 | 9 | 60
  >33-67% | 10 | 10 | 11 | 12 | 17 | 19 | 79
  >67-100% | 4 | 1 | 0 | 1 | 0 | 0 | 6
  NA | 0 | 0 | 1 | 1 | 0 | 0 | 2
Epithelial defect [Mean (Inter-Quartile Range); unit: mm] | 3.2 [2.3 to 3.9] | 3 [2.2 to 3.5] | 3.0 [2.4 to 4.0] | 3.9 [2.6 to 4.5] | 3.5 [2.2 to 4.5] | 3.4 [3.0 to 4.7] | 3.2 [2.5 to 4.2]
Duration of symptoms [Median (Inter-Quartile Range); unit: days] | 3 [2 to 5] | 4 [3 to 14] | 5 [4 to 10] | 7 [3 to 7] | 5 [3 to 10] | 4 [3 to 9] | 5 [3 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Microbiological Cure on Repeat Culture
Description: Corneal scraping of the ulcer will be performed and directly inoculated on to sheep's blood agar, chocolate agar, potato dextrose agar or Sabouraud's agar for bacterial and fungal culture. Microbiological cure is defined as no growth of bacteria or fungus on these media.
Time Frame: 4 to 24 hours after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Bacterial Ulcer Control | Bacterial Ulcer Cross-linking | Fungal Ulcer Control With Natamycin | Fungal Ulcer Cross-linking Plus Natamycin | Fungal Ulcer Control With Amphotericin | Fungal Ulcer Cross-linking Plus Amphotericin
Number analyzed (Participants) | 19 | 16 | 26 | 26 | 27 | 26
Participants
  Culture negative | 5 | 5 | 17 | 14 | 15 | 13
  Culture positive | 14 | 11 | 9 | 12 | 12 | 13

2. Secondary Outcome: Best Spectacle-corrected Visual Acuity
Description: Best corrected visual acuity will be measured at baseline for both eyes using the standard ETDRS chart light box at the 4- and 1-meter test distances. In the case that the patient reads less than 10 letters at 4 meters, move the patient or the chart to a distance of 1 meter from the patient.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: logMar
Arm/Group | Bacterial Ulcer Control | Bacterial Ulcer Cross-linking | Fungal Ulcer Control With Natamycin | Fungal Ulcer Cross-linking Plus Natamycin | Fungal Ulcer Control With Amphotericin | Fungal Ulcer Cross-linking Plus Amphotericin
Number analyzed (Participants) | 17 | 16 | 21 | 27 | 27 | 25
logMar | 0.82 [0.62 to 1.4] | 1.32 [0.43 to 1.75] | 0.43 [0.1 to 0.72] | 1 [0.3 to 1.8] | 0.48 [0.2 to 1.7] | 0.8 [0.5 to 1.24]

3. Secondary Outcome: Scar Size
Description: Study clinician will measure infiltrate or scar size using a standardized protocol with the slit lamp biomicroscope. The geometric mean of the scar size will be measured by recording the horizontal and vertical diameter.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- Fungal Ulcer Cross-linking Plus Amphotericin: tandard of care topical treatment for fungal ulcer with amphotericin plus cross-linking Fungal ulcer cross-linking: Prior to receiving cross-linking, topical amphotericin B or topical natamycin antifungal therapy will be started as per routine at the hospital; a loading dose of amphotericin B or natamycin every 5 minutes x 6 will be followed by dosing every 30 minutes. Amphotericin B and natamycin are routinely used therapies for fungal keratitis at Aravind Eye Hospital.
  For those subjects randomized to receive collagen cross-linking, the procedure will be performed as per the routine at the hospital (UV-X machine; strict aseptic precautions; corneal epithelium debrided and 0.1% riboflavin applied for 30 minutes, then UV-A radiation applied for 30 minutes at 370nm with 3mW/cm2). Corneal cross-linking is a routine procedure performed by Aravind Eye Hospital for infectious keratitis.
Arm/Group | Bacterial Ulcer Control | Bacterial Ulcer Cross-linking | Fungal Ulcer Control With Natamycin | Fungal Ulcer Cross-linking Plus Natamycin | Fungal Ulcer Control With Amphotericin | Fungal Ulcer Cross-linking Plus Amphotericin
Number analyzed (Participants) | 19 | 17 | 26 | 27 | 30 | 28
mm | 3.5 [2.7 to 4.0] | 3.0 [2.24 to 4.0] | 3.0 [2.5 to 3.5] | 3.9 [2.6 to 4.5] | 3.5 [2.7 to 4.5] | 3.1 [2.8 to 5.0]

4. Secondary Outcome: Adverse Events Including Rate of Perforation/Need for Therapeutic Penetrating Keratoplasty
Description: Adverse events include glaucoma, endophthalmitis, medication reaction, perforation including treatment by therapeutic penetrating keratoplasty.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Bacterial Ulcer Control | Bacterial Ulcer Cross-linking | Fungal Ulcer Control With Natamycin | Fungal Ulcer Cross-linking Plus Natamycin | Fungal Ulcer Control With Amphotericin | Fungal Ulcer Cross-linking Plus Amphotericin
Number analyzed (Participants) | 19 | 17 | 26 | 27 | 30 | 28
participants
  Perforation | 1 | 0 | 2 | 1 | 4 | 3
  Therapeutic penetrating keratoplasty | 3 | 1 | 5 | 5 | 5 | 3
  Endophthalmitis | 0 | 0 | 0 | 0 | 1 | 0
  Median tarsorrhaphy | 0 | 0 | 0 | 0 | 0 | 1

5. Other Pre Specified Outcome: Vision Related Quality of Life
Description: Mobility subscale: As measured by the Indian Visual Function Questionnaire (IVFQ) which records quality of life on a scale of 0 to 100 with 100 representing the best quality of life.
Time Frame: 3 months
Population: These data were exploratory in nature, we did not collect the data.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Fungal Ulcer Cross-linking Plus Natamycin: Standard of care topical treatment for fungal ulcer with either natamycin plus cross-linking
  Fungal ulcer cross-linking: Prior to receiving cross-linking, topical natamycin antifungal therapy will be started as per routine at the hospital; a loading dose of natamycin every 5 minutes x 6 will be followed by dosing every 30 minutes. Natamycin are routinely used therapies for fungal keratitis at Aravind Eye Hospital.
  For those subjects randomized to receive collagen cross-linking, the procedure will be performed as per the routine at the hospital (UV-X machine; strict aseptic precautions; corneal epithelium debrided and 0.1% riboflavin applied for 30 minutes, then UV-A radiation applied for 30 minutes at 370nm with 3mW/cm2). Corneal cross-linking is a routine procedure performed by Aravind Eye Hospital for infectious keratitis.
- Fungal Ulcer Cross-linking Plus Amphotericin: Standard of care topical treatment for fungal ulcer with amphotericin plus cross-linking
  Fungal ulcer cross-linking: Prior to receiving cross-linking, topical amphotericin B will be started as per routine at the hospital; a loading dose of amphotericin B every 5 minutes x 6 will be followed by dosing every 30 minutes. Amphotericin B are routinely used therapies for fungal keratitis at Aravind Eye Hospital.
  For those subjects randomized to receive collagen cross-linking, the procedure will be performed as per the routine at the hospital (UV-X machine; strict aseptic precautions; corneal epithelium debrided and 0.1% riboflavin applied for 30 minutes, then UV-A radiation applied for 30 minutes at 370nm with 3mW/cm2). Corneal cross-linking is a routine procedure performed by Aravind Eye Hospital for infectious keratitis.
Arm/Group | Bacterial Ulcer Control | Bacterial Ulcer Cross-linking | Fungal Ulcer Cross-linking Plus Natamycin | Fungal Ulcer Control With Natamycin | Fungal Ulcer Control With Amphotericin | Fungal Ulcer Cross-linking Plus Amphotericin
Number analyzed (Participants) | 0 | 0 | 27 | 26 | 30 | 28
score on a scale |  |  | 89.6 [71.9 to 100] | 91.7 [75 to 100] | 95.8 [72.9 to 100] | 89.6 [71.9 to 100]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events were systematically assessed at every study visit.
Arm/Group | Bacterial Ulcer Control | Bacterial Ulcer Cross-linking | Fungal Ulcer Control With Natamycin | Fungal Ulcer Cross-linking Plus Natamycin | Fungal Ulcer Control With Amphotericin | Fungal Ulcer Cross-linking Plus Amphotericin
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17 | 0/26 | 0/27 | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 4/19 | 1/17 | 7/26 | 6/27 | 10/30 | 6/28
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17 | 0/26 | 0/27 | 0/30 | 1/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bacterial Ulcer Control (N=19) | Bacterial Ulcer Cross-linking (N=17) | Fungal Ulcer Control With Natamycin (N=26) | Fungal Ulcer Cross-linking Plus Natamycin (N=27) | Fungal Ulcer Control With Amphotericin (N=30) | Fungal Ulcer Cross-linking Plus Amphotericin (N=28)
Perforation (Eye disorders) | 1 | 0 | 2 | 1 | 4 | 3
Therapeutic penetrating keratoplasty (Eye disorders) | 3 | 1 | 5 | 5 | 5 | 3
Endophthalmitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bacterial Ulcer Control (N=19) | Bacterial Ulcer Cross-linking (N=17) | Fungal Ulcer Control With Natamycin (N=26) | Fungal Ulcer Cross-linking Plus Natamycin (N=27) | Fungal Ulcer Control With Amphotericin (N=30) | Fungal Ulcer Cross-linking Plus Amphotericin (N=28)
Median tarsorrhaphy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT02570321/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT02570321/SAP_001.pdf
  • Informed Consent Form (2016-05-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT02570321/ICF_002.pdf